CLINICAL TRIAL: NCT05251207
Title: The Role of Gut Microbiota Metabolite, Trimethylamine N-oxide, in the Insulin Resistance Development
Brief Title: Plasma Trimethylamine N-oxide Elevation Induced by L-carnitine Supplementation and Insulin Resistance
Acronym: MR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Robert Olek, Principal Investigator, Poznan University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020/39/O/NZ7/01790
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Carnitine; Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- carnitine (Experimental): 2 grams of L-carnitine per day for 12 weeks
  Interventions: Dietary Supplement: L-carnitine; Behavioral: Change of the circadian cycle
- leucine (Placebo Comparator): 2 grams of L-leucine per day for 12 weeks
  Interventions: Dietary Supplement: L-leucine; Behavioral: Change of the circadian cycle
- modified circadian cycle (Experimental): no sleep at night for four consecutive days (enabling sleep between 8:00 and 17:00).
  Interventions: Dietary Supplement: L-carnitine; Dietary Supplement: L-leucine
- normal circadian cycle (Active Comparator): sleep at night for four consecutive days
  Interventions: Dietary Supplement: L-carnitine; Dietary Supplement: L-leucine

INTERVENTIONS:
Dietary Supplement: L-carnitine — L-carnitine-L-tartrate
  Arms: carnitine; modified circadian cycle; normal circadian cycle
Dietary Supplement: L-leucine — L-leucine
  Arms: leucine; modified circadian cycle; normal circadian cycle
Behavioral: Change of the circadian cycle — Reducing sleep at night for four consecutive days (enabling sleep between 8:00 and 17:00)
  Arms: carnitine; leucine

SUMMARY:
The primary aims of the current study:

* using L-carnitine supplementation modulate the level of plasma trimethylamine N-oxide to assess its effect on circulating cytokines related to diabetes and metabolic syndrome;
* using simulated night-shift work intervention as a stress factor, explore the effect of circulating metabolites on insulin sensitivity

The secondary aim is to evaluate the effect of carnitine supplementation on gut microbiome composition.

DETAILED DESCRIPTION:
Subjects will be randomly divided in two groups: supplemented by L-carnitine 2g/day for 12 weeks, and placebo group receiving leucine in identical gelatine capsules.

Subjects who successfully complete the protocol will be divided into four subgroups - two with a changed circadian cycle and two controls (supplemented and placebo). Subgroups with a changed daily cycle will be able to sleep between 8:00 and 17:00 for four consecutive days, while during the night they will stay active in the laboratory. The oral glucose tolerance test (OGTT) will be performed before and after the circadian cycle modification. Glucose levels will be monitored by FreeStyle Libre Sensor. Moreover, the activity of the participants will be monitored by wearable activity trackers.

Before supplementation, as well as before circadian cycle modification and after finishing the whole experimental procedure, fasting blood samples will be collected for determination of plasma trimethylamine N-oxide (TMAO), trimethylamine (TMA), carnitine (free and acyl derivatives), protein markers of diabetes and inflammation.

Moreover, the stool samples will be collected before and after 12 weeks of supplementation, to determine the composition of the gut microbiome. In addition diet of participants will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers,
* must be able to swallow tablets

Exclusion Criteria:

* smokers,
* cardiovascular disease
* liver disease
* kidney disease
* gastrointestinal disorders (including stomach ulcers and erosions)
* diabetes

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Circulating microbiome metabolites | 13 weeks
  Determination of plasma trimethylamine and trimethylamine N-oxide using ultra performance liquid chromatography - tandem mass spectrometer (UPLC-MS/MS) method
Circulating carnitine metabolites | 13 weeks
  Determination of plasma free, total, and acyl-L-carnitines using ultra performance liquid chromatography - tandem mass spectrometer (UPLC-MS/MS) method
Circulating diabetes biomarkers | 13 weeks
  insulin, C-peptide, ghrelin, leptin, resistin using enzyme-linked immunosorbent assay
Circulating inflammatory biomarkers | 13 weeks
  tumor necrosis factor, C-reactive protein using enzyme-linked immunosorbent assay
Oral Glucose Tolerance Test | 1 week
  The subjects will consume 75 g of glucose solution drink within a 5-minute time frame. The glucose level will be continuously monitored with the FreeStyle Libre Sensor.

SECONDARY OUTCOMES:
gut microbiome composition | 13 weeks
  16 S rRNA sequencing will be used to analyze the gut microbiome in the stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Robert Olek, PhD, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Akademia Wychowania Fizycznego, Poznan, Poland

REFERENCES:
- [Background] Samulak JJ, Sawicka AK, Hartmane D, Grinberga S, Pugovics O, Lysiak-Szydlowska W, Olek RA. L-Carnitine Supplementation Increases Trimethylamine-N-Oxide but not Markers of Atherosclerosis in Healthy Aged Women. Ann Nutr Metab. 2019;74(1):11-17. doi: 10.1159/000495037. Epub 2018 Nov 28. PMID 30485835
- [Background] Bescos R, Boden MJ, Jackson ML, Trewin AJ, Marin EC, Levinger I, Garnham A, Hiam DS, Falcao-Tebas F, Conte F, Owens JA, Kennaway DJ, McConell GK. Four days of simulated shift work reduces insulin sensitivity in humans. Acta Physiol (Oxf). 2018 Jun;223(2):e13039. doi: 10.1111/apha.13039. Epub 2018 Feb 12. PMID 29356345